CLINICAL TRIAL: NCT01003847
Title: Differential Metabolic Effects of Fenofibrate and Fatty Acid
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gachon University Gil Medical Center (Other)
Responsible Party: Dr. Koh, Gachon University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GMC-200911
Record Dates: First submitted 2009-10-28; First posted 2009-10-29 (Estimated); Last update posted 2011-05-10 (Estimated); Status verified 2010-10

CONDITIONS: Hypertriglyceridemia
Keywords: Insulin resistance
MeSH Terms: conditions — Hypertriglyceridemia; Insulin Resistance | interventions — Fenofibrate; Fatty Acids

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- fenofibrate (Active Comparator)
  Interventions: Drug: fenofibrate, fatty acid, placebo
- fatty acid (Active Comparator): drug
  Interventions: Drug: fenofibrate, fatty acid, placebo
- Placebo (Active Comparator)
  Interventions: Drug: fenofibrate, fatty acid, placebo

INTERVENTIONS:
Drug: fenofibrate, fatty acid, placebo — fenofibrate 160 mg, fatty acids 2 gm, placeob 8 weeks of treatment

SUMMARY:
The investigators hypothesize that fenofibrate and fatty acid may have different metabolic effects in hypertriglyceridemic patients

ELIGIBILITY:
Inclusion Criteria:

* hypertriglyceridemia

Exclusion Criteria:

* Overt liver disease Chronic renal failure Hypothyroidism Myopathy Uncontrolled diabetes Severe hypertension

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2009-11; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
flow-mediated dilation | 8 weeks of treatment

SECONDARY OUTCOMES:
insulin resistance | 8 weeks of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Gil Medical Center, Incheon, South Korea